CLINICAL TRIAL: NCT00982553
Title: A Prospective, Open-label, Three Phase Pharmacokinetic Study, to Assess the Pharmacokinetic Profile and Safety of Raltegravir 400 mg Twice Daily and Ribavirin 800 mg Once Daily, When Dosed Separately and Together in Healthy Volunteers
Brief Title: The Raltegravir and Ribavirin Pharmacokinetics (PK) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-010005-36; 2009-010005-36 (EudraCT Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections
Keywords: Healthy Volunteers
MeSH Terms: conditions — HIV Infections | interventions — Ribavirin; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1_ribavirin (Experimental): Treatment with Single dose ribavirin (800 mg) administered on day 1
  Interventions: Drug: Ribavirin
- Phase2_raltegravir (Experimental): Treatment with Raltegravir (400 mg twice daily) administered from days 15-19
  Interventions: Drug: Raltegravir
- Phase3_ribavirin+raltegravir (Experimental): Treatment with Ribavirin (800 mg) and Raltegravir (400 mg) administered day 20
  Interventions: Drug: Ribavirin; Drug: Raltegravir

INTERVENTIONS:
Drug: Ribavirin — 800mg once daily
  Other Names: Copegus
  Arms: Phase 1_ribavirin; Phase3_ribavirin+raltegravir
Drug: Raltegravir — 400mg twice daily
  Arms: Phase2_raltegravir; Phase3_ribavirin+raltegravir

SUMMARY:
The purpose of this study is to look at levels of both a new anti-HIV drug called raltegravir and an existing anti-hepatitis C drug called ribavirin to see if they affect the blood levels of each other when given separately and together. This is a phase I, open-label, prospective, three phase, pharmacokinetic study.

DETAILED DESCRIPTION:
Phase I (study day 1 - 14):

* 14 healthy volunteers with a documented negative HIV-1 antibody test during screening procedures will be enrolled.
* On day 1, fasted subjects will be administered ribavirin 800 mg without food (witnessed dosing). This will be followed be a 12 hour detailed pharmacokinetic assessment; blood sampling drawn at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 and 12 hours.
* This will be followed by a wash-out period.
* As steady state pharmacokinetics of ribavirin are not reached for several weeks, single dosing pharmacokinetics will be assessed in this study

Phase II (study days 15 - 19):

* On day 15, subjects will commence raltegravir 400 mg twice daily. Subjects will attend for safety visits and witnessed dosing during this phase.
* Day 19 - after 4 days of dosing when steady state pharmacokinetics has been reached, subjects will attend for a 12 hour detailed pharmacokinetic visit where following witnessed administration of raltegravir 400 mg without food, blood sampling will be drawn at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post dose for the assessment of raltegravir plasma exposure.

Phase III (study day 20):

• Subjects will be administered raltegravir 400 mg and ribavirin 800 mg without food. This will be followed by a 12 hour detailed pharmacokinetic assessment with blood sampling drawn at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.
* Male or non-pregnant, non-lactating female.
* Between 18 to 60 years, inclusive.
* Subjects in good health upon medical history, physical exam, and laboratory testing and body mass index below 32.
* Female subjects who are heterosexually active and of childbearing potential (i.e., not surgically sterile or at least two years post menopausal) must practice contraception as follows from screening through completion of the study including 180 days following last dose of study drug:

  * barrier contraceptives (condom, diaphragm with spermicide)
  * oral combined contraceptive pill, implant or injectable hormonal contraceptive PLUS a barrier contraceptive
  * Intrauterine device (IUD) or intrauterine system (IUS) PLUS a barrier contraceptive (or a partner who has been vasectomized for at least six months).
* Female subjects of childbearing potential must have a negative urine pregnancy test.
* Male subjects who are heterosexually active must use two forms of barrier contraception (e.g., condom with spermicide) during heterosexual intercourse, from screening through completion of the study including 180 days following last dose of study drug.
* Have no serologic evidence of HIV infection.
* Have no serologic evidence of active hepatitis B virus infection evidenced by negative hepatitis B surface antigen and no serologic evidence of hepatitis C virus infection through antibody testing.
* Have screening laboratory results (haematology, chemistry) that fall within the normal range of the central laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance.

Exclusion Criteria:

* Any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include any active clinically significant renal, cardiac, hepatic, pulmonary, vascular, metabolic (thyroid disorders, adrenal disease), immunodeficiency disorders, active infection, or malignancy.
* Have a body mass index (BMI) greater than 32
* Previous participation in an investigational trial involving administration of any investigational compound within 1 month prior to the study screening.
* Clinically relevant alcohol or drug use (positive screening drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
* Any medication taken listed in Prior and Concomitant Medication section including over-the-counter medications and herbal products within 21 days of commencing study drug dosing with the exception of vitamins and/or paracetamol and/or hormonal contraceptives including the combined oral contraceptive pill, Depo-Provera and the Mirena intrauterine system. When a concomitant medication is necessary, this will be reviewed by the Investigator and if not contraindicated, may be continued at the same dose and frequency during the study period.
* History of drug sensitivity or drug allergy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MB BH, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ashby J, Garvey L, Erlwein OW, Lamba H, Weston R, Legg K, Latch N, McClure MO, Dickinson L, D'Avolio A, Back D, Winston A. Pharmacokinetic and safety profile of raltegravir and ribavirin, when dosed separately and together, in healthy volunteers. J Antimicrob Chemother. 2011 Jun;66(6):1340-5. doi: 10.1093/jac/dkr093. Epub 2011 Mar 15. PMID 21406434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Recruitment was between 24/09/2009 and 29/10/2009.
  * 14 subjects were enrolled.
  * The study took place at a specialist research unit at an National Health Service (NHS) hospital.
Pre-assignment Details: * Subjects were healthy volunteers.
  * There was a 21 day washout for any prescribed and 7 days for over the counter medication before enrolment.
  * The subjects were permitted to take paracetamol during the study but all others were excluded for the duration of the trial.
Groups:
- All Subjects: All subjects received the same study therapy as follows:
  Day 1 Ribavirin single dose 800 mg oral followed by intensive PK monitoring. Day 2 - 14 washout phase Day 15 - 18 raltegravir 400 mg twice daily followed by by intensive PK monitoring on day 18.
  Day 19 raltegravir 400 mg plus ribavirin 800 mg by intensive PK monitoring.
Period: Phase1
Arm/Group | All Subjects
Started | 14
Completed | 14
Not Completed | 0
Period: Phase2
Arm/Group | All Subjects
Started | 14
Completed | 14
Not Completed | 0
Period: Phase3
Arm/Group | All Subjects
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14

OUTCOME MEASURES:

1. Primary Outcome: Ribavirin Maximum Plasma Concentration
Description: Pharmacokinetic analyses of blood samples
Time Frame: Day 20
Population: Per protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Phase1_ribavirin: Single dose ribavirin 800mg administered on day 1
- Phase3_ribovarin and Raltegravir: Single dose ribavirin 800mg and raltegravir 400mg at day 20
Arm/Group | Phase1_ribavirin | Phase3_ribovarin and Raltegravir
Number analyzed (Participants) | 14 | 14
ng/mL | 630.09 [490.91 to 808.54] | 496.71 [407.38 to 605.76]
Statistical Analysis 1: Comparison: Phase1_ribavirin vs Phase3_ribovarin and Raltegravir; Test type: Superiority; Geometric mean ratios = 0.79, 95% CI 2-sided [0.62 to 1.00]

2. Primary Outcome: Raltegravir Maximum Plasma Concentration
Time Frame: Day 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Phase2_Raltegravir: Raltegravir 400 mg twice daily on day 15-19
- Phase3_ribovarin and Raltegravir: On day 20 single dose of both ribavirin and raltegravir administered together
Arm/Group | Phase2_Raltegravir | Phase3_ribovarin and Raltegravir
Number analyzed (Participants) | 14 | 14
ng/mL | 2227.41 [1489.36 to 3331.19] | 2591.19 [1778.28 to 3774.85]
Statistical Analysis 1: Comparison: Phase2_Raltegravir vs Phase3_ribovarin and Raltegravir; Test type: Superiority; Geometric mean ratios = 1.16, 95% CI 2-sided [0.73 to 1.86]

3. Primary Outcome: Ribavirin Minimum Plasma Concentration
Description: Ribavirin minimum plasma concentration by pharmacokinetic analyses
Time Frame: Day 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Phase3_ribovarin and Raltegravir: Onn day 20 single dose of both ribavirin and raltegravir administered together
Arm/Group | Phase1_Ribavirin | Phase3_ribovarin and Raltegravir
Number analyzed (Participants) | 14 | 14
ng/mL | 184.71 [148.59 to 229.61] | 186.98 [157.83 to 221.56]
Statistical Analysis 1: Comparison: Phase1_Ribavirin vs Phase3_ribovarin and Raltegravir; Test type: Superiority; Geometric mean ratios = 1.01, 95% CI 2-sided [0.87 to 1.18]

4. Primary Outcome: Raltegravir Minimum Plasma Concentrations
Description: Raltegravir minimum plasma concentrations by pharmacokinetic analyses
Time Frame: Day 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Phase2_Raltegravir | Phase3_ribovarin and Raltegravir
Number analyzed (Participants) | 14 | 14
ng/mL | 83.97 [45.64 to 154.45] | 68.91 [40.74 to 116.55]
Statistical Analysis 1: Comparison: Phase2_Raltegravir vs Phase3_ribovarin and Raltegravir; Test type: Superiority; Geometric mean ratios = 0.82, 95% CI 2-sided [0.36 to 1.85]

ADVERSE EVENTS:
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No